CLINICAL TRIAL: NCT00953459
Title: Phase II Study of Sunitinib (SU011248) in Patients With Small Cell Lung Cancer Who Are Either Chemo-naïve (Extensive Disease) or Have a "Sensitive" Relapse
Brief Title: Sunitinib Malate in Treating Patients With Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poorly recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08061; EU-20910; 2006-002485-19 (EudraCT Number)
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Sunitinib; Fluorodeoxyglucose F18

INTERVENTIONS:
Drug: sunitinib malate
Other: laboratory biomarker analysis
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib malate works in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the therapeutic activity of sunitinib malate in patients with either chemonaïve extensive stage or sensitive relapsed small cell lung cancer.

Secondary

* To characterize the safety of sunitinib malate in these patients.

Tertiary

* To determine the potential of FDG-PET-scan to serve as a surrogate marker of response for the antiangiogenic activity of the compound.

OUTLINE: This is a multicenter study. Patients are stratified according to disease stage (chemonaïve extensive stage vs sensitive relapse at least 3 months after stopping chemotherapy).

Patients receive oral sunitinib malate once daily for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients undergo fludeoxyglucose F 18 positron emission tomography of the chest at week 4. Blood samples and bronchial washings and brushings may be collected at baseline and at 4 and 8 weeks after start of therapy for further analysis.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer

  * Chemotherapy naïve (extensive stage) OR sensitive relapse (> 3 months since induction therapy) disease
* Measurable disease, as defined by RECIST criteria
* No brain metastases as assessed by CT scan or MRI performed < 1 week before treatment

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* AST and ALT ≤ 2.5 x upper limit of normal (ULN) (≤ 5 x ULN if liver function abnormalities are due to underlying malignancy)
* Total serum bilirubin ≤ 1.5 x ULN
* Serum albumin ≥ 3.0 g/dL
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study treatment
* No spinal cord compression, carcinomatous meningitis, or leptomeningeal disease
* No myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus within the past 6 months
* No NCI CTCAE grade 3 hemorrhage within the past 4 weeks
* No hypertension (> 150/100 mm Hg) that cannot be controlled with standard antihypertensive agents
* No ongoing cardiac dysrhythmias of grade ≥ 2, atrial fibrillation of any grade, or QTc interval > 450 msec for males or > 470 msec for females
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study drug administration or may interfere with the interpretation of study results, and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy, surgery, or investigational agents
* At least 1 month since prior radiotherapy except for palliative radiotherapy to non-target lesions
* No prior treatment with sunitinib malate (SU011248) or other receptor tyrosine kinase inhibitors
* No concurrent treatment with steroids
* No concurrent treatment with a drug having proarrhythmic potential (i.e., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide)
* More than 7 and 12 days and no concurrent potent CYP3A4 inhibitors and inducers, respectively
* Concurrent coumarin-derivative anticoagulants, such as warfarin (Coumadin®) up to 2 mg daily are permitted for prophylaxis of thrombosis
* No other concurrent anticancer treatments, including chemotherapy, immunotherapy, targeted agents, hormonal cancer therapy, radiation therapy, or experimental treatments

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Disease control rate (percentage of patients with complete response, partial response, or stable disease) 8 weeks after beginning treatment according to RECIST criteria

SECONDARY OUTCOMES:
Response rate every 4 weeks according to RECIST criteria
Duration of progression-free survival
Duration of response
Duration of survival
Toxicity according to NCI CTCAE version 3.0
Accuracy of FDG-PET scan as a potential early surrogate marker of antiangiogenic activity for response

CONTACTS AND LOCATIONS:
Overall Officials: Egbert F. Smit, MD, Principal Investigator — Free University Medical Center
Locations (1):
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands